CLINICAL TRIAL: NCT01681030
Title: A Randomized, Controlled, Comparative Phase II Study Evaluating the Safety and Effectiveness of EVARREST™ Fibrin Sealant Patch as an Adjunct to Hemostasis During Cardiovascular Surgery
Brief Title: The Fibrin Pad Cardiovascular Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 400-12-002
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Results first posted 2018-03-07 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fibrin Tissue Adhesive; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EVARREST™ (Experimental): EVARREST™ Fibrin Sealant Patch is a sterile bio-absorbable combination product consisting of two constituent parts- a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin).
  Interventions: Biological: EVARREST™
- Topical hemostat (Active Comparator): Equine collagen with Human Fibrinogen and Human Thrombin
  Interventions: Biological: Topical hemostat
- Standard of Care (Active Comparator): SoC is a composite of techniques/methods typically used by the surgeon to control bleeding after conventional methods (i.e. suture, ligation, cautery) are ineffective or impractical.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Biological: EVARREST™ — EVARREST™ Fibrin Sealant Patch is a sterile bio-absorbable combination product consisting of two constituent parts- a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin).
  Arms: EVARREST™
Biological: Topical hemostat — Equine collagen with Human Fibrinogen and Human Thrombin
  Arms: Topical hemostat
Other: Standard of Care — SoC is a composite of techniques/methods typically used by the surgeon to control bleeding after conventional methods (i.e. suture, ligation, cautery) are ineffective or impractical.
  Arms: Standard of Care

SUMMARY:
This is a three-arm, randomized multicenter study evaluating the safety and effectiveness of EVARREST™ Fibrin Sealant Patch in controlling mild to moderate vascular anastomosis suture line bleeding in cardiovascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years of age, requiring an elective or urgent, open aortic surgical procedure utilizing cardiopulmonary bypass;
* Subjects must be willing to participate in the study and provide written informed consent.

Exclusion Criteria:

* Subjects with known intolerance to blood products or to one of the components of the study product or unwilling to receive blood products;
* Exposure to another investigational drug or device in a clinical trial within 30 days prior to surgery or anticipated in the 30 day follow up period after surgery.
* Female subjects who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2013-08-01 (Actual); Study Completion 2013-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Riebman, MD, Study Director — Ethicon, Inc.
Locations (6):
- United States (6):
  - Clinical Investigation Site #5, Indianapolis, Indiana
  - Clinical Investigation Site #6, Kansas City, Missouri
  - Clinical Investigation Site #4, Camden, New Jersey
  - Clinical Investigation Site #1, Paterson, New Jersey
  - Clinical Investigation Site #3, New York, New York
  - Clinical Investigation Site #2, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from September 17, 2012 through September 3, 2013 at hospitals and medical centers throughout the United States.
Groups:
- EVARREST Fibrin Sealant Patch: EVARREST® Fibrin Sealant Patch is a sterile bio-absorbable combination product consisting of two constituent parts - a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin.
- Topical Hemostat: Equine collagen sponge with Human Fibrinogen and Human Thrombin
- Standard of Care (SoC): SoC is a composite of techniques/methods typically used by the surgeon to control bleeding after conventional methods (i.e. suture, ligation, cautery) are ineffective or impractical.
Period: Overall Study
Arm/Group | EVARREST Fibrin Sealant Patch | Topical Hemostat | Standard of Care (SoC)
Started | 13 | 18 | 11
Completed | 13 | 18 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data was summarized for Intent to Treat (ITT) Set, which included all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | EVARREST Fibrin Sealant Patch | Topical Hemostat | Standard of Care (SoC) | Total
Number analyzed (Participants) | 13 | 18 | 11 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 56.0 (15.1) | 59.8 (12.9) | 60.5 (15.4) | 58.8 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 9
  Male | 9 | 15 | 9 | 33
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 0 | 1 | 1
  Black or African American | 2 | 0 | 2 | 4
  White/Caucasian | 9 | 11 | 6 | 26
  Hispanic or Latino | 2 | 7 | 2 | 11
BMI Category [Number; unit: Participant] — Underweight: < 18.5 kg/m^2, Normal weight: 18.5 - <25 kg/m^2 , Overweight: 25 - <30 kg/m^2, Obese: 30 - <40 kg/m^2, Morbidly obese: 40 kg/m^2 or more
  Participant
    Normal | 5 | 7 | 4 | 16
    Overweight | 3 | 5 | 2 | 10
    Obese | 3 | 5 | 4 | 12
    Morbidly obese | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Hemostasis at the Target Bleeding Site (TBS) at 3 Minutes Following Treatment Application.
Description: Number of subjects achieving hemostasis at the Target Bleeding Site (TBS) at 3 minutes following treatment application, with no re-bleeding at the TBS any time prior to the initiation of final chest wall closur
Time Frame: Intraoperative, 3 minutes following treatment application
Measure: Count of Participants; unit: Participants
Arm/Group | EVARREST Fibrin Sealant Patch | Topical Hemostat | Standard of Care (SoC)
Number analyzed (Participants) | 13 | 18 | 11
Participants | 12 | 6 | 5
Statistical Analysis 1: Comparison: EVARREST Fibrin Sealant Patch; Test type: Superiority or Other; Proportion = 0.923, 95% CI 2-sided [0.640 to 0.998] — CI for EVARREST Group
Statistical Analysis 2: Comparison: Topical Hemostat; Test type: Superiority or Other; Proportion = 0.333, 95% CI 2-sided [0.133 to 0.590] — CI for Topical Hemostat group
Statistical Analysis 3: Comparison: Standard of Care (SoC); Test type: Superiority or Other; Proportion = 0.455, 95% CI 2-sided [0.167 to 0.766] — CI for Standard of Care group

2. Secondary Outcome: Hemostasis at the Target Bleeding Site (TBS) at 6 Minutes Following Treatment Application
Description: The number of subjects achieving hemostatic success at 6 minutes following treatment application.
Time Frame: Intraoperative, 6 minutes following treatment application
Measure: Count of Participants; unit: Participants
Arm/Group | EVARREST Fibrin Sealant Patch | Topical Hemostat | Standard of Care (SoC)
Number analyzed (Participants) | 13 | 18 | 11
Participants | 12 | 11 | 7

3. Secondary Outcome: Hemostasis at the Target Bleeding Site (TBS) at 10 Minutes Following Treatment Application
Description: Number of subjects achieving hemostatic success at 10 minutes following treatment application.
Time Frame: Intraoperative, 10 minutes following treatment application
Measure: Count of Participants; unit: Participants
Arm/Group | EVARREST Fibrin Sealant Patch | Topical Hemostat | Standard of Care (SoC)
Number analyzed (Participants) | 13 | 18 | 11
Participants | 12 | 12 | 8

4. Secondary Outcome: Bleeding at the Target Bleeding Site (TBS) Requiring Additional Treatment
Description: The number of subjects who, after the initial establishment of TBS hemostasis at 3 minutes, had re-bleeding requiring treatment
Time Frame: Intra-operative, prior initiation of final chest wall closure. Safety Issue:
Population: Subjects who established TBS hemostasis at 3 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | EVARREST Fibrin Sealant Patch | Topical Hemostat | Standard of Care (SoC)
Number analyzed (Participants) | 12 | 11 | 5
Participants | 0 | 5 | 0

5. Secondary Outcome: Number of Participants With Adverse Events Potentially Related to Thrombotic Events
Description: The number of subjects with an adverse event potentially related to a thrombotic event
Time Frame: 30 days (+ 14 days) following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | EVARREST Fibrin Sealant Patch | Topical Hemostat | Standard of Care (SoC)
Number analyzed (Participants) | 13 | 18 | 11
Participants | 0 | 2 | 2

ADVERSE EVENTS:
Time Frame: From surgical procedure through the 30 day follow-up (+/- 14 days)
Arm/Group | EVARREST Fibrin Sealant Patch | Topical Hemostat | Standard of Care (SoC)
Serious Adverse Events (participants affected / at risk) | 3/13 | 10/18 | 6/11
Other Adverse Events (participants affected / at risk) | 13/13 | 18/18 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EVARREST Fibrin Sealant Patch (N=13) | Topical Hemostat (N=18) | Standard of Care (SoC) (N=11)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
RENAL FAILURE (Renal and urinary disorders) | 0 | 1 | 0
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 2 | 0 | 0
SPINAL CORD ISCHAEMIA (Nervous system disorders) | 0 | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 2 | 0
PNEUMONIA (Infections and infestations) | 0 | 1 | 0
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 | 0 | 0
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 | 0 | 1
SINUS BRADYCARDIA (Cardiac disorders) | 0 | 1 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 0 | 1
CARDIAC TAMPONADE (Cardiac disorders) | 0 | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 0 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 | 3 | 1
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 2 | 1
COAGULOPATHY (Blood and lymphatic system disorders) | 0 | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EVARREST Fibrin Sealant Patch (N=13) | Topical Hemostat (N=18) | Standard of Care (SoC) (N=11)
HYPOTENSION (Vascular disorders) | 3 | 7 | 2
HYPERTENSION (Vascular disorders) | 0 | 1 | 0
HAEMATOMA (Vascular disorders) | 0 | 1 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 2 | 2
THORACIC CAVITY DRAINAGE (Surgical and medical procedures) | 1 | 0 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 5
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
CHRONIC OBSTRUCTIVE PULMONARY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 4
URINARY RETENTION (Renal and urinary disorders) | 0 | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 1 | 1 | 0
DELIRIUM (Psychiatric disorders) | 0 | 1 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 2 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 2
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 2 | 0 | 0
AGITATION (Psychiatric disorders) | 0 | 1 | 0
SPINAL CORD ISCHAEMIA (Nervous system disorders) | 0 | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
FRACTURE MALUNION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 1 | 0
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 2
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 2 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 2 | 0
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 | 1 | 0
ACIDOSIS (Metabolism and nutrition disorders) | 0 | 1 | 1
RED BLOOD CELL COUNT DECREASED (Investigations) | 1 | 0 | 0
PLATELET COUNT DECREASED (Investigations) | 0 | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0 | 0
HAEMATOCRIT DECREASED (Investigations) | 1 | 0 | 0
BLOOD FIBRINOGEN INCREASED (Investigations) | 0 | 0 | 1
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 | 1 | 0
TRANSFUSION-RELATED ACUTE LUNG INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 | 1 | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 2 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 1 | 0 | 0
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 1 | 1
FUNGAL INFECTION (Infections and infestations) | 0 | 0 | 1
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 1 | 0
BACTERAEMIA (Infections and infestations) | 0 | 0 | 1
PYREXIA (General disorders) | 2 | 0 | 2
OEDEMA PERIPHERAL (General disorders) | 0 | 3 | 2
OEDEMA (General disorders) | 0 | 3 | 2
HYPOTHERMIA (General disorders) | 0 | 1 | 0
FATIGUE (General disorders) | 0 | 1 | 0
EFFUSION (General disorders) | 0 | 1 | 1
CHEST PAIN (General disorders) | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 1 | 0
PEPTIC ULCER (Gastrointestinal disorders) | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 4 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 1 | 0
FLATULENCE (Gastrointestinal disorders) | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 2 | 3 | 3
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 | 0 | 1
TACHYCARDIA (Cardiac disorders) | 0 | 2 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0
SINUS BRADYCARDIA (Cardiac disorders) | 0 | 1 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 0 | 1
CARDIAC TAMPONADE (Cardiac disorders) | 0 | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1 | 1
CARDIAC FAILURE (Cardiac disorders) | 1 | 0 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 0 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 | 3 | 1
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 | 1 | 0
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 5 | 3
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 4 | 2
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 2 | 0
COAGULOPATHY (Blood and lymphatic system disorders) | 1 | 1 | 2
ANAEMIA (Blood and lymphatic system disorders) | 3 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days